CLINICAL TRIAL: NCT06351631
Title: A Multicenter, Open-Label, Extension Study Evaluating the Safety and Efficacy of Bomedemstat for the Treatment of Participants Enrolled in a Prior Bomedemstat Clinical Study
Brief Title: A Study to Evaluate Safety and Efficacy of Bomedemstat (MK-3543-017)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3543-017; 2023-506996-89-00 (Registry Identifier: EU CT); U1111-1294-8621 (Registry Identifier: UTN); MK-3543-017 (Other: MSD)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Thrombocythemia, Essential; Primary Myelofibrosis; Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Polycythemia Vera
MeSH Terms: conditions — Thrombocythemia, Essential; Primary Myelofibrosis; Polycythemia Vera | interventions — bomedemstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bomedemstat (Experimental): Participants will receive oral capsules of bomedemstat once daily for up to 10 years, with the starting dose as the same dose that the participant was on at the time of transition from the feeder study.
  Interventions: Drug: Bomedemstat

INTERVENTIONS:
Drug: Bomedemstat — 10, 15, 20, and 50 mg oral capsules
  Other Names: MK-3543; IMG-7289

SUMMARY:
The primary purpose of the study is to transition participants into an extension study to collect long-term safety and efficacy data. The study will include participants who are safely tolerating bomedemstat, receiving clinical benefit from its use in estimation of the investigator, and have shown the following criteria:

* Participants from the IMG-7289-202/MK-3543-005 (NCT05223920) study must have received at least 6 months of treatment with bomedemstat;
* Essential thrombocythemia (ET) and polycythemia vera (PV) participants from studies other than IMG-7289-202/MK-3543-005 must have achieved confirmed hematologic remission.

No hypothesis testing will be conducted in this study.

ELIGIBILITY:
Inclusion Criteria:

* Is from a bomedemstat study sponsored by Imago BioSciences, Inc. (a subsidiary of Merck & Co., Inc.) or MSD, and established by the Sponsor as MK-3543-017 ready
* Has received at least 6 months of treatment with bomedemstat in the IMG-7289-202/MK-3543-005 study, while safely tolerating bomedemstat, and receiving clinical benefit from its use in the estimation of the investigator
* ET and PV participants from established feeder studies other than IMG-7289- 202/MK-3543-005 must have achieved confirmed hematologic remission, must be safely tolerating bomedemstat, and must be receiving clinical benefit from its use in the estimation of the investigator
* Is not currently on a dose hold
* Participant must be able to swallow oral medication and follow instructions for at-home dosing of bomedemstat

Exclusion Criteria:

* Has received prohibited concomitant medications
* Ongoing or planned participation in another investigational study
* Has noncompliance in prior bomedemstat study receiving <90% of assigned doses excluding suspensions or holds as assigned by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2034-12-04 (Estimated); Study Completion 2034-12-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with one or more adverse events (AEs) | Up to ~10 years
  An AE is any undesirable physical, psychological or behavioral effect experienced by a patient during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. This includes any untoward signs or symptoms experienced by the patient from the time of first dose with bomedemstat under this protocol until completion of the study. The percentage of participants with AEs will be presented.
Percentage of participants who discontinued study treatment due to an AE | Up to ~10 years
  An AE is any undesirable physical, psychological or behavioral effect experienced by a patient during participation in an investigational study, in conjunction with the use of the drug or biologic, whether or not product-related. This includes any untoward signs or symptoms experienced by the patient from the time of first dose with bomedemstat under this protocol until completion of the study. The percentage of participants who discontinued study treatment due to an AE will be presented.

SECONDARY OUTCOMES:
For participants with ET or PV: Duration of clinicohematologic response | Up to ~10 years
  For participants who showed durable clinicohematologic response (DCHR) in their feeder studies, duration of clinicohematologic response is defined as the time from the first documented evidence of confirmed reduction of platelet and white blood cell (WBC) count until confirmed increase of platelet and WBC counts to above acceptable threshold, thrombotic or major hemorrhagic events or disease progression to myelofibrosis (MF), myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). The duration of clinicohematologic response will be reported.
For participants with ET or PV: Duration of hematologic remission | Up to ~10 years
  For participants who showed confirmed hematologic remission in their feeder studies, duration of hematologic remission is defined as the time from the first documented evidence of confirmed reduction of platelet and WBC count until confirmed increase of platelet and WBC counts to above acceptable threshold. The duration of hematologic remission will be reported.
For participants with ET or PV: Percentage of participants with transformation to MF or MDS/AML | Up to ~10 years
  Disease Progression is defined as the transformation to post-ET myelofibrosis (ET participants only), post-PV myelofibrosis (PV participants only), spleen volume increase ≥25% (MF participants only), myelodysplastic syndrome, or acute myeloid leukemia as assessed by the investigator. The percentage of participants with transformation to MF or MDS/AML will be reported.
For participants with MF: Percentage of participants with worsening of splenomegaly or transformation to MDS/AML | Up to ~10 years
  Spleen volume will be assessed by magnetic resonance imaging (MRI) (or computed tomography [CT] where applicable) at pre-specified timepoints. The percentage of participants with worsening of splenomegaly or transformation to MDS/AML will be reported.
For participants with MF, ET, or PV: Percentage of participants with thrombotic events | Up to ~10 years
  Thrombotic events are defined as: new or recurrent acute myocardial infarction; unstable angina; stroke; transient ischemic attack (TIA); deep venous thrombosis (DVT); pulmonary embolism (PE); thrombotic digital ischemia; other thrombotic events such as peripheral limb ischemia or Budd-Chiari syndrome that are assessed to be due to underlying PV; other vascular occlusive events such as symptoms of cardiac, abdominal or peripheral limb ischemia supported by objective evidence of vessel disease and/or ischemia. The percentage of participants with thrombotic events will be presented.
For participants with MF, ET, or PV: Percentage of participants with major hemorrhagic events | Up to ~10 years
  Hemorrhagic events are defined as: Major Bleeding (MB) Events such as fatal bleeding, and/or symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of 2 or more units of whole blood or red cells; Clinically Relevant Non-Major Bleeding (CRNMB) Events Leading to hospitalization or increased level of care or clinically important, prompting a face-to-face medical evaluation. The percentage of participants with major hemorrhagic events will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (21):
- United States (4):
  - University of Michigan ( Site 6000), Ann Arbor, Michigan
  - DUHS Duke Blood Cancer Center ( Site 6005), Durham, North Carolina
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 6007), Columbus, Ohio
  - UPMC Hillman Cancer Center ( Site 6004), Pittsburgh, Pennsylvania
- Australia (6):
  - Royal Prince Alfred Hospital ( Site 1003), Camperdown, New South Wales
  - Royal North Shore Hospital ( Site 1001), St Leonards, New South Wales
  - Sunshine Coast Hematology and Oncology Clinic ( Site 1006), Buderim, Queensland
  - Gold Coast University Hospital-Cancer and Blood Disorders Clinical Trial Team ( Site 1002), Southport, Queensland
  - Royal Adelaide Hospital-Haematology Clinical Trials Unit ( Site 1000), Adelaide, South Australia
  - Monash Health ( Site 1004), Clayton, Victoria
- Queen Mary Hospital ( Site 1601), Hksar, Hong Kong
- Italy (4):
  - Azienda Ospedaliero-Universitaria SS. Antonio e Biagio e Cesare Arrigo ( Site 2703), Alessandria, Ancona
  - Azienda Ospedaliera Universitaria Careggi ( Site 2700), Florence, Tuscany
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 2702), Bologna
  - Ospedale di Circolo e Fondazione Macchi Varese ( Site 2701), Varese
- New Zealand (2):
  - North Shore Hospital-Department of Haematology ( Site 1401), Auckland
  - Aotearoa Clinical Trials ( Site 1400), Auckland
- United Kingdom (4):
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital ( Site 3402), London, Hammersmith and Fulham
  - Boston Pilgrim Hospital ( Site 3403), Boston, Lincolnshire
  - University College London Hospital ( Site 3400), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust ( Site 3401), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26338&tenant=MT_MSD_9011